CLINICAL TRIAL: NCT00563992
Title: Pharmacotherapy of High-Risk Bipolar Disorder
Brief Title: Effectiveness of Lithium and Valproate in Treating High-Risk Bipolar Disorder
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: #4973R; R01MH059710 (NIH); DSIR 83-ATP
Record Dates: First submitted 2007-11-23; First posted 2007-11-27 (Estimated); Last update posted 2012-05-01 (Estimated); Status verified 2012-04

CONDITIONS: Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder | interventions — Lithium; Valproic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Participants will take lithium for 12 months
  Interventions: Drug: Lithium
- 2 (Experimental): Participants will take valproate for 12 months
  Interventions: Drug: Valproic acid

INTERVENTIONS:
Drug: Lithium — Participants may also be required to take the antidepressant paroxetine and/or the medication olanzapine for a portion of the study.
  Arms: 1
Drug: Valproic acid — Participants may also be required to take the antidepressant paroxetine and/or the medication olanzapine for a portion of the study.
  Other Names: Sodium valproate or valproic acid (Depakote)
  Arms: 2

SUMMARY:
This study will evaluate the effectiveness of two different mood stabilizing medications, lithium and valproate, in treating people with bipolar disorder and suicidal behavior.

DETAILED DESCRIPTION:
Bipolar disorder, also called manic-depressive illness, is a brain disorder that causes dramatic changes in a person's mood and energy. Bipolar disorder normally forms in late adolescence or early adulthood and requires treatment for the rest of a person's life. People with bipolar disorder undergo periods of extreme happiness and extreme sadness, known as episodes of mania and depression. Symptoms of mania can include increased energy, euphoric moods, mind racing, aggressive behavior, substance abuse, and poor decision making. Symptoms of depression can include persistent feelings of anxiety, guilt, or hopelessness; irregular sleep and appetite patterns; lethargy; disinterest in previously enjoyed activities; excessive irritability and restlessness; and inability to concentrate. Some people with bipolar disorder also become suicidal. Suicidal behaviors are more likely to occur at the onset of the illness, making it vital to recognize and treat the disorder early on. Current treatments include mood stabilizing medications and psychotherapy. This study will evaluate the effectiveness of two different mood stabilizing medications, lithium and valproate, in treating people with bipolar disorder and suicidal behavior.

Participants in this double-blind study will be randomly assigned to take one of two medications, either lithium or valproate. In the first 2 to 6 months, depending on clinical condition, participants may also be required to take the antidepressant paroxetine and/or the medication olanzapine. Participants will attend regular visits to a psychiatrist or a psychologist at the Neuroscience Clinic. A blood sample will be taken at each visit to monitor medication blood levels. Participants will also undergo periodic routine laboratory and urine tests to assure their safety.

If the psychiatrist feels improvement has occurred by the end of the 2- to 6-month period, participants will be gradually taken off paroxetine and/or olanzapine over a 2-week period. They will then continue taking the assigned lithium or valproate for the remainder of the study. If the psychiatrist feels the condition has worsened, participants will be prescribed new medications as needed. These medications include other antidepressants (bupropion or venlafaxine) or other antimanic or antipsychotic drugs (perphenazine or haloperidol). Once these participants have achieved at least 2 weeks of normal moods, they will be gradually taken off all other prescribed medications and will remain taking the assigned lithium or valproate. Participants who do not achieve at least 2 weeks of normal moods will stop study participation but will still be offered clinical treatment. The remaining participants taking only lithium or valproate will continue their regular visits with a psychiatrist for the last 6 months of the study. The entire study will last 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Current major depressive episode or mixed episode
* Bipolar disorder
* History of suicidal behavior

Exclusion Criteria:

* Requires detoxification from alcohol or other substances
* Blood pressure greater than 160/90 mm Hg
* Active medical problems
* Requires long-term antipsychotic maintenance
* Becomes manic on mood stabilizers and antidepressants
* Contraindication to the use of lithium 1 or valproate (including failure to respond)
* Failure to respond to adequate trials of paroxetine, bupropion, and venlafaxine in the 2 years prior to study entry
* Failure to respond to adequate trials of olanzapine, haloperidol, and perphenazine in the 2 years prior to study entry
* Unable or unwilling to consent to treatment
* Pregnant or lactating

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2001-01; Primary Completion 2008-09 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Severity of depression and mania by SADS-C (Schedule for Affective Disorders and Schizophrenia, Change) and LIFE (Longitudinal Interval Follow-up Evaluation) | Measured between Months 2 and 6 and at Month 12
Suicide history form and Scale for Suicidal Ideation | Measured between Months 2 and 6 and at Month 12

CONTACTS AND LOCATIONS:
Overall Officials: Maria A. Oquendo, MD, Principal Investigator — Columbia University
Locations (1):
- New York State Psychiatric Institute/Columbia University, New York, New York, United States